CLINICAL TRIAL: NCT06212063
Title: Aim High: Readiness & Meeting the Standards in Military Pre-Recruits
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Tiffany Stewart, Professor, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PBRC 2023-074
Record Dates: First submitted 2023-12-19; First posted 2024-01-18 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aim High Program (Experimental): Integrated physical and mental optimization training program used as tool for young individuals readying themselves to join the military
  Interventions: Behavioral: Cadet Health

INTERVENTIONS:
Behavioral: Cadet Health — Integrated physical and mental optimization training program used as tool for young individuals readying themselves to join the military

SUMMARY:
The primary objective of the proposed study is to complete a comprehensive needs assessment of the Louisiana National Guard (LANG) Youth Challenge Program (YCP) in the YCP leadership and junior cadet population related to nutrition, fitness, sleep, and mental health and resilience. Results of this needs assessment will further inform the development of the intervention skills training program.

The secondary objective of this work is to provide a scalable, integrated physical and mental optimization training program that would be integrated into relevant systems and maintained over time as a core tool for young individuals readying themselves to join the Army. The program would include an environmental intervention approach as well as nutrition, physical activity, sleep, and stress reduction/positive coping guidance.

ELIGIBILITY:
Inclusion Criteria:

* Must be either staff, cadre, or cadets in the YCP program.

Exclusion Criteria:

* Not staff, cadre, or cadets in the YCP program.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Height | 16 Months
  Height for BMI calculations
Weight | 16 Months
  Weight for BMI calculations
Body Fat | 16 Months
  Body Fat % to determine change pre/post program
Depression | 16 Months
  Patient Health Questionnaire for Adolescents (PHQ-8A) to determine change pre/post program; Scores range from 0 to 24, with a higher score meaning higher levels of depressive symptomology
Anxiety | 16 Months
  Generalized Anxiety Disorder Screener (GAD7) to determine change pre/post program; Score range from 0 to 21, with higher scores meaning higher levels of anxiety
Body Esteem | 16 Months
  Body Esteem Scale for Adolescent and Adults (BESAA) to determine change pre/post program; scores range from 0 to 92, with higher scores meaning higher levels of body esteem.
Coping | 16 Months
  Brief COPE; 14 facets of coping skills are assessed and can be consolidated into approach and avoidant coping strategies, with higher scores indicating higher levels of that particular coping strategy
Perceived Stress | 16 Months
  Perceived Stress Scale (PSS); Scores range from 0 to 40, with higher scores meaning higher levels of perceived stress
Eating Competence | 16 Months
  Eating Competence Scale (ecSatter); Scores range from 0 to 48, with higher scores meaning better competence around eating behaviors

SECONDARY OUTCOMES:
Knowledge & Attitudes | 16 Months
  General Questionnaire to assess uptake of knowledge presented in the program; Higher scores will indicate higher levels of understanding of key program concepts
Program Satisfaction | 16 Months
  Questionnaire to determine program acceptability; Higher scores indicate higher satisfaction with program content and delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No